CLINICAL TRIAL: NCT01640834
Title: Pilot Study of the Effects of LY2409021 in Patients With Type 1 Diabetes Mellitus
Brief Title: Study of LY2409021 in Participants With Type 1 Diabetes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 14576; I1R-MC-GLBR (Other: Eli Lilly and Company); 2011-006178-19 (EudraCT Number)
Record Dates: First submitted 2012-07-12; First posted 2012-07-16 (Estimated); Results first posted 2018-10-29 (Actual); Last update posted 2018-10-29 (Actual); Status verified 2018-03

CONDITIONS: Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — adomeglivant; Glucagon

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 100 mg LY2409021 (Experimental): LY2409021: 100 milligrams (mg), 1 capsule, administered as a single oral dose on Day 2.
  Placebo: 2 capsules, administered as a single oral dose on Day 2.
  Glucagon: 1 mg administered via intramuscular injection on Day 3.
  Interventions: Drug: LY2409021; Drug: Placebo; Drug: Glucagon
- 300 mg LY2409021 (Experimental): LY2409021: 300 milligrams (mg), 3 capsules (3 X 100-mg capsules), administered as a single oral dose on Day 2.
  Glucagon: 1 mg administered via intramuscular injection on Day 3.
  Interventions: Drug: LY2409021; Drug: Glucagon
- Placebo (Placebo Comparator): Placebo: 3 capsules administered as a single oral dose on Day 2.
  Glucagon: 1 milligram (mg) administered via intramuscular injection on Day 3.
  Interventions: Drug: Placebo; Drug: Glucagon

INTERVENTIONS:
Drug: LY2409021 — Administered orally
  Arms: 100 mg LY2409021; 300 mg LY2409021
Drug: Placebo — Administered orally
  Arms: 100 mg LY2409021; Placebo
Drug: Glucagon — Administered via intramuscular injection

SUMMARY:
This study involves taking a single dose of 100 milligrams (mg) or 300 mg LY2409021 or placebo (an inactive medicine) taken as up to 3 capsules by mouth. The study will evaluate if this drug will reduce the amount of insulin a type 1 diabetic needs over 24 hours. This study includes a 7-day hospitalization period at the clinical research unit (CRU) and will involve screening within 30 days of the start of the study as well as telephone consultations within 5 days after discharge from the CRU.

ELIGIBILITY:
Inclusion Criteria:

* Have had type 1 diabetes mellitus (T1DM) based on the World Health Organization classification for at least 1 year and have a daily insulin dose ≤1.5 international units (IU) per kilogram (kg) of body weight
* Have a glycated hemoglobin A1c (HbA1c) of no greater than 9.0% as measured at screening
* Have a body mass index (BMI) ≥19.0 and ≤35.0 kilograms per meter squared (kg/m^2)
* Have given written informed consent approved by Lilly

Exclusion Criteria:

* Received any oral or injectable medication intended for the treatment of diabetes mellitus other than insulins in the 3 months prior to screening
* Have had more than 1 episode of severe hypoglycemia within 3 months prior to entry into the study, or are currently diagnosed as having hypoglycemia unawareness
* Are pregnant or intend to become pregnant during the course of the study
* Women who are breastfeeding
* Have a history of stroke, myocardial infarction, heart failure, unstable angina, or a coronary revascularization procedure within 6 months of screening
* Have fasting triglycerides >500 milligrams per deciliter (mg/dL) (5.65 millimoles per liter [mmol/L])
* Have obvious clinical signs, symptoms, or laboratory evidence of liver disease (alanine transaminase [ALT] or aspartate transaminase [AST] greater than 2 times the upper limit of normal at screening)
* Have a history of renal transplantation or are currently receiving renal dialysis or have a screening creatinine >2.0 mg/dL (177 micromoles per liter [μmol/L])
* Have had any other disease, illness, or condition (including known diabetic autonomic neuropathy, drug or alcohol abuse, or psychiatric disorder) within the 6 months prior to screening that precludes the participant from following and completing the study or could increase their risk for hypoglycemia, according to the investigator's judgment
* Are currently enrolled in, have completed, or have discontinued within the last 30 days from a clinical trial involving an off-label use of an investigational drug or device, or are concurrently enrolled in any other type of medical research judged not to be scientifically or medically compatible with this study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2012-07; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Neuss, Germany

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 100 mg LY2409021 | 300 mg LY2409021 | Placebo
Started | 8 | 8 | 4
Received at Least 1 Dose of Study Drug | 8 | 8 | 4
Completed | 8 | 8 | 4
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | 100 mg LY2409021 | 300 mg LY2409021 | Placebo | Total
Number analyzed (Participants) | 8 | 8 | 4 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.6 (12.8) | 47.1 (5.7) | 43.3 (10.6) | 43.0 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 8 | 8 | 4 | 20
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 8 | 8 | 4 | 20
Region of Enrollment [Count of Participants; unit: Participants]
  Germany | 8 | 8 | 4 | 20

OUTCOME MEASURES:

1. Primary Outcome: Pharmacodynamics: Change From Baseline to Day 2 in 24-hour Insulin Dose
Description: The mean absolute change in total insulin dose over 24 hours (Day 2, 24-hour insulin dose - Day 1, 24-hour insulin dose) is reported.
Time Frame: Baseline (Day 1), Day 2
Population: All participants who received a dose of LY2409021 or placebo and had evaluable 24-hour insulin data.
Measure: Mean (Standard Deviation); unit: insulin units
Arm/Group | 100 mg LY2409021 | 300 mg LY2409021 | Placebo
Number analyzed (Participants) | 8 | 8 | 4
insulin units | 1.85 (7.15) | 0.80 (9.63) | 7.69 (2.99)
Statistical Analysis 1: Comparison: 100 mg LY2409021; The mean change on Day 2 from Day 1 in the 24-hour insulin dose for the placebo group was subtracted from each participant's change on Day 2 from Day 1 in the 24-hour insulin dose. This placebo adjusted 24-hour insulin dose was compared within the 100-mg LY2409021 dose group using a 1 sample t-test; Test type: Superiority or Other; p = 0.0542, t-test, 1 sided; Mean Difference (Net) = -5.84, 95% CI 2-sided [-11.82 to 0.14]
Statistical Analysis 2: Comparison: 300 mg LY2409021; The mean change on Day 2 from Day 1 in the 24-hour insulin dose for the placebo group was subtracted from each participant's change on Day 2 from Day 1 in the 24-hour insulin dose. This placebo adjusted 24-hour insulin dose was compared within the 300-mg LY2409021 dose group; Test type: Superiority or Other; p = 0.0826, t-test, 1 sided; Mean Difference (Net) = -6.89, 95% CI 2-sided [-14.95 to 1.16]

2. Secondary Outcome: Pharmacodynamics: Percentage Change From Baseline to Day 2 in 24-hour Insulin
Description: The percentage change in total insulin dose over 24 hours (Day 2, 24-hour insulin dose - Day 1, 24-hour insulin dose) is reported.
Time Frame: Baseline (Day 1), Day 2
Population: All participants who received a dose of LY2409021 or placebo and had evaluable 24-hour insulin data.
Measure: Mean (Standard Deviation); unit: percentage of insulin units
Arm/Group | 100 mg LY2409021 | 300 mg LY2409021 | Placebo
Number analyzed (Participants) | 8 | 8 | 4
percentage of insulin units | 5.71 (19.90) | 3.12 (18.34) | 22.75 (22.20)
Statistical Analysis 1: Comparison: 100 mg LY2409021; Analysis was performed using the percent change in insulin dose, which takes into account absolute differences in individual insulin doses. The mean percent change on Day 2 from Day 1 in the 24-hour insulin dose for the placebo group was subtracted from each participant's percent change on Day 2 from Day 1 in the 24-hour insulin dose. This placebo adjusted 24-hour insulin dose was compared within the 100-mg LY2409021 dose group using a 1 sample t-test; Test type: Superiority or Other; p = 0.0460, t-test, 1 sided; Mean Difference (Net) = -17.0, 95% CI 2-sided [-33.7 to -0.4]
Statistical Analysis 2: Comparison: 300 mg LY2409021; Analysis was performed using the percent change in insulin dose, which takes into account absolute differences in individual insulin doses. The mean percent change on Day 2 from Day 1 in the 24-hour insulin dose for the placebo group was subtracted from each participant's percent change on Day 2 from Day 1 in the 24-hour insulin dose. This placebo adjusted 24-hour insulin dose was compared within the 300-mg LY2409021 dose group using a 1 sample t-test; Test type: Superiority or Other; p = 0.0192, t-test, 1 sided; Mean Difference (Net) = -19.6, 95% CI 2-sided [-35.0 to -4.3]

3. Secondary Outcome: Pharmacokinetics: Maximum Concentration (Cmax) of LY2409021
Time Frame: Predose (Day 2) through 120 hours postdose (Day 7)
Population: All participants who received a dose of LY2409021 and had evaluable pharmacokinetic data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter
Arm/Group | 100 mg LY2409021 | 300 mg LY2409021
Number analyzed (Participants) | 8 | 8
nanograms per milliliter | 2620 (23) | 6090 (23)

4. Secondary Outcome: Pharmacokinetics: Area Under the Concentration Curve (AUC) of LY2409021
Description: Exposure in terms of AUC of LY2409021 from time 0 extrapolated to infinity (AUCinf) is reported.
Time Frame: Predose (Day 2) through 120 hours postdose (Day 7)
Population: All participants who received a dose of LY2409021 and had evaluable pharmacokinetic data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms * hours per milliliter
Groups:
- 100 mg LY2409021: LY2409021: 100 milligrams (mg), capsule, administered as a single oral dose on Day 2.
  Placebo: 2 capsules, administered as a single oral dose on Day 2.
  Glucagon: 1 mg administered via intramuscular injection on Day 3.
- 300 mg LY2409021: LY2409021: 300 milligrams (mg), capsules (3 X 100-mg capsules), administered as a single oral dose on Day 2.
  Glucagon: 1 mg administered via intramuscular injection on Day 3.
Arm/Group | 100 mg LY2409021 | 300 mg LY2409021
Number analyzed (Participants) | 8 | 8
nanograms * hours per milliliter | 209000 (30) | 506000 (22)

5. Secondary Outcome: Pharmacodynamics: Change From Baseline in 24 Hour Insulin Dose During Drug Washout Period
Description: Data were not captured, and, therefore, this outcome measure was not analyzed. Zero participants were included in the analysis.
Time Frame: Baseline (Day 1), Day 3 up to Day 6
Population: This outcome measure was not analyzed.
Arm/Group | 100 mg LY2409021 | 300 mg LY2409021 | Placebo
Number analyzed (Participants) | 0 | 0 | 0

6. Secondary Outcome: Pharmacodynamics: Change From Baseline in 24 Hour Insulin Dose Needed to Maintain Euglycemia
Description: as for outcome 5
Time Frame: Baseline (Day 1), Day 3 up to Day 6
Population: This outcome measure was not analyzed.
Arm/Group | 100 mg LY2409021 | 300 mg LY2409021 | Placebo
Number analyzed (Participants) | 0 | 0 | 0

7. Secondary Outcome: Pharmacodynamics: Maximum Concentration (Cmax) of Glucose Concentration After 1 Milligram (mg) Glucagon Injection on Day 3
Description: The Cmax of glucose following a single dose of glucagon (1 mg) administered via an intramuscular injection is reported.
Time Frame: Day 3
Population: All participants who received a dose of LY2409021 or placebo and had evaluable post-glucagon injection glucose concentration data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: milligrams per deciliter
Arm/Group | 100 mg LY2409021 | 300 mg LY2409021 | Placebo
Number analyzed (Participants) | 8 | 8 | 4
milligrams per deciliter | 154.9 (19) | 141.3 (19) | 201.8 (11)
Statistical Analysis 1: Comparison: 100 mg LY2409021 vs Placebo; Statistical analysis of the effect of LY2409021 treatment on peak glucose concentration after an intramuscular injection of glucagon (1 milligram); Test type: Superiority or Other; p = 0.0187, t-test, 2 sided; Mean Difference (Net) = -46, 95% CI 2-sided [-82 to -9]
Statistical Analysis 2: Comparison: 300 mg LY2409021 vs Placebo; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; p = 0.0048, t-test, 2 sided; Mean Difference (Net) = -59, 95% CI 2-sided [-96 to -23]

8. Secondary Outcome: Pharmacodynamics: Area Under the Glucose Concentration Curve After a Single Dose of Glucagon on Day 3
Description: Area under the glucose concentration curve from time 0 through 2 hours after a single dose of glucagon (1 milligram) administered via an intramuscular injection is reported.
Time Frame: Day 3
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: milligrams * minutes per deciliter
Arm/Group | 100 mg LY2409021 | 300 mg LY2409021 | Placebo
Number analyzed (Participants) | 8 | 8 | 4
milligrams * minutes per deciliter | 15534.3 (21) | 14885.5 (16) | 20189.7 (9)
Statistical Analysis 1: Comparison: 100 mg LY2409021 vs Placebo; Statistical analysis of the effect of LY2409021 treatment on area under the glucose concentration curve from time 0 to 2 hours postdose following an intramuscular injection of glucagon (1 milligram); Test type: Superiority or Other; p = 0.0278, t-test, 2 sided; Mean Difference (Net) = -4423, 95% CI 2-sided [-8256 to -590]
Statistical Analysis 2: Comparison: 300 mg LY2409021 vs Placebo; [analysis description as in outcome 8, analysis 1]; Test type: Superiority or Other; p = 0.0046, t-test, 2 sided; Mean Difference (Net) = -5187, 95% CI 2-sided [-8371 to -2004]

ADVERSE EVENTS:
Arm/Group | 100 mg LY2409021 | 300 mg LY2409021 | Placebo
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/4
Other Adverse Events (participants affected / at risk) | 6/8 | 6/8 | 4/4
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 100 mg LY2409021 (N=8) | 300 mg LY2409021 (N=8) | Placebo (N=4)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Discomfort (General disorders) | 0 (0) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 6 (19) | 6 (13) | 3 (6)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days